CLINICAL TRIAL: NCT03242824
Title: MC167B: Pilot Study Investigating the Utility of 18F-DOPA-PET in the Treatment of Recurrent High-grade Glioma
Brief Title: The Utility of 18F-DOPA-PET in the Treatment of Recurrent High-grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-006072; MC167B (Other: Cancer Center Identifier); NCI-2017-02479 (Other: NCI)
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Results first posted 2022-07-05 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — fluorodopa F 18; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-DOPA PET (Experimental): Patients will receive 18FDOPA-PET for radiation treatment planning
  Interventions: Drug: Fluorine F 18 Fluorodopa; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Fluorine F 18 Fluorodopa — Contrast used in PET
  Other Names: 18F- FDOPA; 3,4-dihydroxy-6-[18F] fluoro-L-phenylalanine
Radiation: Intensity-Modulated Radiation Therapy — Radiation of different intensities are aimed at the tumor from many angles. This type of radiation therapy reduces the damage to healthy tissue near the tumor
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Procedure: Positron Emission Tomography — imaging test
  Other Names: PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography

SUMMARY:
This proposal is for a pilot study comparing volumes of 18F-DOPA-PET avidity with contrast enhancement and T2 FLAIR on MRI. Investigators then plan to compare patterns of failure with target volumes, pre-treatment MRI changes and pre-treatment 18F-DOPA-PET.

ELIGIBILITY:
Inclusion Criteria

* Age > or equal to 18 years
* ECOG PS < or equal to 3
* Histologically confirmed or radiographic evidence of recurrent/progressive glioma.
* History of radiation therapy to the brain for prior diagnosis of glioma
* Planned radiation treatments at Mayo Clinic Rochester
* Provide informed written consent
* Willing to sign consent onto the Mayo Clinic Radiotherapy Patient Outcomes Registry and Biobanking study, IRB number 15-000136 (blood draw optional)
* Willing to return to enrolling institution for follow-up during Active Monitoring Phase of the study.

Exclusion Criteria

* More than one prior course of radiotherapy or prior prescription doses exceeding 60 Gy to re-irradiation target volumes
* Unable to undergo MRI scans with contrast
* Unable to undergo an 18F-DOPA-PET scan (e.g., Parkinson's Disease, taking anti dopaminergic, or dopamine agonist medication or less than 6 half-lives from discontinuance of dopamine agonists.)

Note: Other potentially interfering drugs: amoxapine, amphetamine, benztropine, buproprion, buspirone, cocaine, mazindol, methamphetamine, methylphenidate, norephedrine, phentermine, phenylpropanolamine, selegiline, paroxetine, citalopram, and sertraline). If a patient is on any of these drugs, list which ones on the On-Study form.

-Any of the following:

* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2021-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N Laack, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 registered patient did not proceed to protocol treatment because they were deemed ineligible.
Groups:
- 18F-DOPA PET: Patients will receive 18FDOPA-PET for radiation treatment planning. Fluorine F 18 Fluorodopa: Contrast used in PET. Intensity-Modulated Radiation Therapy: Radiation of different intensities are aimed at the tumor from many angles. This type of radiation therapy reduces the damage to healthy tissue near the tumor. Positron Emission Tomography: imaging test
Period: Overall Study
Arm/Group | 18F-DOPA PET
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18F-DOPA PET
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 53 [38 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Progression-free Survival
Description: measured by reviewing 18F-DOPA-PET and conventional MRI with historical controls
Time Frame: up to 3 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | 18F-DOPA PET
Number analyzed (Participants) | 20
Proportion of participants | 0.85 [0.632 to 0.958]

2. Secondary Outcome: Overall Survival
Description: Overall survival from initial diagnosis: Time from initial diagnosis to death from any cause censoring patients alive at their last follow-up, assessed up to 2 years from date of randomization
Time Frame: From date of diagnosis to date of death from any cause censoring patients alive at their last follow-up; patients assessed for survival up to 2 years from randomization. Diagnosis date occurs prior to randomization by up to 15 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | 18F-DOPA PET
Number analyzed (Participants) | 20
years | 3.7 [2.4 to NA] — Upper limit on 95% confidence interval is not estimable (NE), due to an insufficient number of participants with events.

3. Secondary Outcome: Toxicity, Rate of Grade 3 or Higher Treatment Related to Toxicities
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0. A copy of the CTCAE version 4.0 can be downloaded from the CTEP web site:(http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm)
Time Frame: up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | 18F-DOPA PET
Number analyzed (Participants) | 20
percentage of participants | 40

4. Secondary Outcome: Quality of Life Brief Fatigue Index (BFI) Change From Baseline
Description: Measured by change from baseline to 3 month evaluation in MDA-BFI global fatigue score. Brief fatigue index is a QOL questionnaire with scores ranging from 0, no fatigue, to 10, as bad as you can imagine.
Time Frame: Baseline and 3 months
Population: All patients that entered a baseline and at 3 months.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | 18F-DOPA PET
Number analyzed (Participants) | 19
score on a scale | 0.28 [-0.75 to 0.78]

5. Secondary Outcome: Re-operative Count
Description: Count of patients that receive re-operation post re-irradiation
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-DOPA PET
Number analyzed (Participants) | 20
Participants | 0

6. Secondary Outcome: Quality of Life MDASI-BT Change From Baseline
Description: QOL will be evaluated using the MD Anderson Symptom Inventory Brain Tumor Module (MDASI-BT) and fatigue will be evaluated using the MD Anderson Brief Fatigue Inventory.Measured by change from baseline to 3 month evaluation in MDASI-BT overall symptom distress score. Scores may range from 0 to 10, with 0 being 'Not present' and 10 being 'As bad as imaginable'.
Time Frame: Baseline and 3 months
Population: All treated patients that had available data at baseline and during end of treatment.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | 18F-DOPA PET
Number analyzed (Participants) | 19
score on a scale | -0.15 [-0.84 to 0.53]

ADVERSE EVENTS:
Time Frame: up to 2 years from randomization
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0. A copy of the CTCAE version 4.0 can be downloaded from the CTEP web site:
  (http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm)
Arm/Group | 18F-DOPA PET
All-Cause Mortality (participants affected / at risk) | 15/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-DOPA PET (N=20)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (4)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Optic nerve disorder (Eye disorders) | 2 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 17 (49)
Urinary tract infection (Infections and infestations) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Central nervous system necrosis (Nervous system disorders) | 7 (14)
Cognitive disturbance (Nervous system disorders) | 12 (23)
Dysphasia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (6)
Memory impairment (Nervous system disorders) | 8 (11)
Muscle weakness left-sided (Nervous system disorders) | 1 (1)
Muscle weakness right-sided (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 6 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03242824/Prot_SAP_001.pdf